CLINICAL TRIAL: NCT04139122
Title: A Randomized, Double-Masked, Single-Center, Placebo-Controlled Single and Multiple Ascending Dose Study to Assess Safety, Tolerability, Pharmacokinetics, and Efficacy of SJP-0132 in Subjects With Dry Eye Disease
Brief Title: Safety, PK and Efficacy Study of SJP-0132 in Subjects With Dry Eye Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Senju Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SJP-0132/1-01
Record Dates: First submitted 2019-10-14; First posted 2019-10-25 (Actual); Results first posted 2023-04-20 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-03

CONDITIONS: Dry Eye Disease; Dry Eye Syndrome
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1-4: SJP-0132 (Experimental): Each cohort will receive a single dose of 1 of 4 strengths of SJP-0132
  Interventions: Drug: SJP-0132
- Cohort 1-4: Placebo (Placebo Comparator): Single dose of placebo
  Interventions: Drug: Placebo
- Cohort 5-6: SJP-0132 (Experimental): Cohort 5 SJP-0132 will receive the second maximum acceptable dose from Cohorts 1-4 for 4 weeks. Cohort 6 SJP-0132 will receive the maximum acceptable dose from Cohorts 1-4 for 4 weeks
  Interventions: Drug: SJP-0132
- Cohort 5-6: Placebo (Placebo Comparator): Multiple dose placebo for 4 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SJP-0132 — SJP-0132 is administered as an eye drop
  Arms: Cohort 1-4: SJP-0132; Cohort 5-6: SJP-0132
Drug: Placebo — Placebo is administered as an eye drop
  Arms: Cohort 1-4: Placebo; Cohort 5-6: Placebo

SUMMARY:
This is the first study in humans to evaluate the effectiveness of SJP-0132 in the treatment of dry eye disease. This study will evaluate the safety, tolerability, efficacy, and pharmacokinetics of single- and multiple-dose regimens of SJP-0132 in subjects with dry eye disease

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) within 18.5 to 30.0 kg/m2 (inclusive) and body weight between 45 kg and 100 kg
* Generally healthy as determined by medical history, physical examinations, clinical laboratory examination, and ophthalmologic examinations performed at Screening
* Have a subject reported history of Dry Eye Disease in both eyes for at least 6 months prior to Screening
* Non-smoker or ex-smoker for >12 months

Exclusion Criteria:

* Have clinically significant systemic or ophthalmic disease
* Has a positive serum pregnancy test at Screening or urine pregnancy test
* Have had significant blood loss or have donated or received one or more units (450 mL) of blood or plasma within 30 days before randomization
* Have used or anticipates use of any prescription or over-the-counter medication, including topical medications such as ophthalmic solutions, nasal drops or spray, vitamins, alternative and complementary medicines (including herbal formulations) within 14 days or 5 half-lives (whichever is longer) before randomization or at any time during the study
* Use or anticipates use of prescribed dry eye medications within 28 days prior to randomization or at any time during the study
* Have used or anticipates use CYP3A4 inducers, such as St. John's Wort, within 14 days before randomization or at any time during the study.
* Have consumed red wine, grapefruit or grapefruit juice, Seville oranges, star fruit, or any products containing these items, or any foods that may inhibit CYP3A4, within 48 hours before randomization and throughout the duration of the study
* Have a positive urine alcohol or urine drug test at Screening or Day -1
* Contact lens wearers who cannot discontinue the wear over the trial period
* Have undergone eye surgery (including laser surgery) within the last 12 months or whom the Investigator considers unsuitable
* Have a best corrected visual acuity (BCVA) worse than 20/100 in either eye
* History of permanent punctal occlusion (cautery or laser) or current use of punctal plugs
* Any corneal abnormality or disease which might impact normal tear film spreading
* Active or history of significant corneal disease
* Known allergy or sensitivity to fluorescein, lissamine green or any of the study medications

Other protocol-defined Inclusion/Exclusion Criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2019-10-05 (Actual); Primary Completion 2020-03-03 (Actual); Study Completion 2020-03-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Senju Investigational Site, Cypress, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Single-dose (Cohort 1): 0.03% SJP-0132: Single dose of 0.03% SJP-0132 as Cohort 1
- Single-dose (Cohort 2) : 0.1% SJP-0132: Single dose of 0.1% SJP-0132 as Cohort 2
- Single-dose (Cohort 3) : 0.3% SJP-0132: Single dose of 0.3% SJP-0132 as Cohort 3
- Single-dose (Cohort 4) : 1% SJP-0132: Single dose of 1% SJP-0132 as Cohort 4
- Single-dose (Cohort 1-4) : Placebo: Single dose of placebo as Cohort 1 to 4
- Multiple-dose (Cohort 5) : 0.3% SJP-0132: Multiple dose of 0.3% SJP-0132 for 4 weeks as Cohort 5
- Multiple-dose (Cohort 6) : 1% SJP-0132: Multiple dose of 1% SJP-0132 for 4 weeks as Cohort 6
- Multiple-dose (Cohort 5, 6) : Placebo: Multiple dose for 4 weeks as Cohort 5 and 6
Period: Overall Study
Arm/Group | Single-dose (Cohort 1): 0.03% SJP-0132 | Single-dose (Cohort 2) : 0.1% SJP-0132 | Single-dose (Cohort 3) : 0.3% SJP-0132 | Single-dose (Cohort 4) : 1% SJP-0132 | Single-dose (Cohort 1-4) : Placebo | Multiple-dose (Cohort 5) : 0.3% SJP-0132 | Multiple-dose (Cohort 6) : 1% SJP-0132 | Multiple-dose (Cohort 5, 6) : Placebo
Started | 6 | 6 | 5 | 4 | 8 | 20 | 20 | 20
Completed | 5 | 6 | 5 | 4 | 8 | 20 | 20 | 19
Not Completed | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Single-dose (Cohort 1) : 0.03% SJP-0132: Single dose of 0.03% SJP-0132 as Cohort 1
- Total: Total of all reporting groups
Arm/Group | Single-dose (Cohort 1) : 0.03% SJP-0132 | Single-dose (Cohort 2) : 0.1% SJP-0132 | Single-dose (Cohort 3) : 0.3% SJP-0132 | Single-dose (Cohort 4) : 1% SJP-0132 | Single-dose (Cohort 1-4) : Placebo | Multiple-dose (Cohort 5) : 0.3% SJP-0132 | Multiple-dose (Cohort 6) : 1% SJP-0132 | Multiple-dose (Cohort 5, 6) : Placebo | Total
Number analyzed (Participants) | 6 | 6 | 5 | 4 | 8 | 20 | 20 | 20 | 89
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.8 (5.64) | 34.8 (7.78) | 35.0 (6.82) | 35.8 (11.87) | 33.0 (6.72) | 46.1 (14.34) | 34.9 (8.07) | 39.7 (11.74) | 37.9 (11.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 3 | 0 | 6 | 13 | 8 | 13 | 50
  Male | 3 | 2 | 2 | 4 | 2 | 7 | 12 | 7 | 39
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 4 | 3 | 2 | 2 | 4 | 14 | 12 | 10 | 51
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Black or African American | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  White | 2 | 3 | 3 | 2 | 2 | 6 | 8 | 10 | 36
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 5 | 4 | 8 | 20 | 20 | 20 | 89
BMI [Mean (Standard Deviation); unit: Kg/m^2] | 24.675 (3.8471) | 23.882 (4.0167) | 24.144 (3.6329) | 24.593 (3.5238) | 23.303 (3.1095) | 23.596 (2.967) | 25.513 (2.9228) | 24.407 (2.7066) | 24.35 (3.0727)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events by Severity in Each Cohort
Description: Number of participants with adverse events by severity are summarize in each cohort. Adverse events are reported as Treatment-Emergent Adverse Events (TEAEs), which are defined as any event not present before exposure to the study drug or any event already presented that worsened in either intensity or frequency after exposure to the study drug.
Time Frame: Day 2 for cohort 1-4, Day 29 for cohort 5-6
Population: Safety set
Measure: Count of Participants; unit: Participants
Groups:
- Multiple-dose (Cohort 5, 6) : Placebo: Multiple dose of placebo for 4 weeks as Cohort 5 and 6
Arm/Group | Single-dose (Cohort 1) : 0.03% SJP-0132 | Single-dose (Cohort 2) : 0.1% SJP-0132 | Single-dose (Cohort 3) : 0.3% SJP-0132 | Single-dose (Cohort 4) : 1% SJP-0132 | Single-dose (Cohort 1-4) : Placebo | Multiple-dose (Cohort 5) : 0.3% SJP-0132 | Multiple-dose (Cohort 6) : 1% SJP-0132 | Multiple-dose (Cohort 5, 6) : Placebo
Number analyzed (Participants) | 6 | 6 | 5 | 4 | 8 | 20 | 20 | 20
Participants
  Mild | 0 | 0 | 2 | 0 | 0 | 1 | 5 | 7
  Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Subjects With Abnormal Changes in Laboratory Parameters, Vital Signs, and/or Physical and Ophthalmologic Observations in Each Cohort
Description: Clinical laboratory parameters include hematology, clinical chemistry, urinalysis, and serology. Vital signs include diastolic blood pressure, systolic blood pressure, heart rate, respiratory rate, and body temperature. Ophthalmologic observations include examination of visual acuity, slit lamp biomicroscopy, Schirmer I, intraocular pressure, and ophthalmoscopy.
Time Frame: Day 2 for cohort 1-4, Day 29 for cohort 5-6
Population: Safety Set
Measure: Count of Participants; unit: Participants
Groups:
- Single-dose (Cohort 1):0.03% SJP-0132: Single dose of 0.03% SJP-0132 as Cohort 1
Arm/Group | Single-dose (Cohort 1):0.03% SJP-0132 | Single-dose (Cohort 2) : 0.1% SJP-0132 | Single-dose (Cohort 3) : 0.3% SJP-0132 | Single-dose (Cohort 4) : 1% SJP-0132 | Single-dose (Cohort 1-4) : Placebo | Multiple-dose (Cohort 5) : 0.3% SJP-0132 | Multiple-dose (Cohort 6) : 1% SJP-0132 | Multiple-dose (Cohort 5, 6) : Placebo
Number analyzed (Participants) | 6 | 6 | 5 | 4 | 8 | 20 | 20 | 20
Participants
  Laboratory parameters | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Vital signs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Physical observations | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 4
  Ophthalmologic observations | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Maximum Plasma Concentration (Cmax)
Description: The results are from the maximum plasma concentration (Cmax) on Day 1. The blood for pharmacokinetics assessment was collected at 0, 0.25, 0.5, 1, 2, 4, 8, and 12 hours after dosing on Day 1 for Cohorts 1 to 4. The blood for pharmacokinetics assessment was collected at 0, 0.25, 0.5, 1, 2, and 4 hours after dosing on Day 1 for Cohorts 5 and 6.
Time Frame: Day 1
Population: Pharmacokinetic Set
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Single-dose (Cohort 2):0.1% SJP-0132: Single dose of 0.1% SJP-0132 as Cohort 2
- Single-dose (Cohort 3):0.3% SJP-0132: Single dose of 0.3% SJP-0132 as Cohort 3
- Single-dose (Cohort 4):1% SJP-0132: Single dose of 1% SJP-0132 as Cohort 4
- Multiple-dose (Cohort 5):0.3% SJP-0132: Multiple dose of 0.3% SJP-0132 for 4 weeks as Cohort 5
- Multiple-dose (Cohort 6):1% SJP-0132: Multiple dose of 1% SJP-0132 for 4 weeks as Cohort 6
Arm/Group | Single-dose (Cohort 1):0.03% SJP-0132 | Single-dose (Cohort 2):0.1% SJP-0132 | Single-dose (Cohort 3):0.3% SJP-0132 | Single-dose (Cohort 4):1% SJP-0132 | Multiple-dose (Cohort 5):0.3% SJP-0132 | Multiple-dose (Cohort 6):1% SJP-0132
Number analyzed (Participants) | 6 | 6 | 5 | 4 | 12 | 12
ng/mL | 0.03773 (0.015911) | 0.12940 (0.095403) | 0.10228 (0.063893) | 0.69275 (0.293932) | 0.14077 (0.106705) | 0.63273 (0.804411)

4. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time 0 to Time of the Last Quantifiable Concentration (AUC0-last)
Description: Area under the plasma concentration-time curves (AUCs) for Cohorts 1 to 4 were calculated using the plasma collected at 0, 0.25, 0.5, 1, 2, 4, 8, and 12 hours after dosing on Day 1, and those for Cohorts 5 and 6 were calculated using the plasma collected at 0, 0.25, 0.5, 1, 2, and 4 hours after dosing on Day 1.
Time Frame: Day 1
Population: Pharmacokinetic Set
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Single-dose (Cohort 1):0.03% SJP-0132 | Single-dose (Cohort 2):0.1% SJP-0132 | Single-dose (Cohort 3):0.3% SJP-0132 | Single-dose (Cohort 4):1% SJP-0132 | Multiple-dose (Cohort 5):0.3% SJP-0132 | Multiple-dose (Cohort 6):1% SJP-0132
Number analyzed (Participants) | 6 | 6 | 5 | 4 | 12 | 12
hr*ng/mL | 0.28671 (0.158116) | 1.02449 (0.827814) | 0.85442 (0.462688) | 5.15571 (2.537673) | 0.32305 (0.178608) | 1.14604 (1.024450)

5. Primary Outcome: Accumulation Ratio (Rac) After Multiple Dosing
Description: Plasma were collected at 0, 0.25, 0.5, 1, 2, and 4 hours after dosing on Day 1, pre-dose on Day 2, Day 4 and Day 8. Accumulation ratios calculated as (predose plasma concentration [Ctrough] on Day 4) / (Ctrough on Day 2) and (Ctrough on Day 8) / (Ctrough on Day 2)
Time Frame: Day 2, 4, 8
Population: Pharmacokinetic Set
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Multiple-dose (Cohort 5):0.3% SJP-0132 | Multiple-dose (Cohort 6):1% SJP-0132
Number analyzed (Participants) | 12 | 12
Ratio
  Rac Day 4/Day 2 | 1.75758 (0.705735) | 1.67083 (0.812324)
  Rac Day 8/Day 2 | 2.84759 (1.858905) | 2.79157 (1.676501)

6. Primary Outcome: Change From Baseline in Eye Dryness Symptom (VAS) at 4hour on Day 29
Description: Visual analog scale (VAS): "0" mean none, and "100" mean the worst imaginable for the symptom question.
Time Frame: Day 29
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Multiple-dose (Cohort 5, 6):Placebo: Multiple dose of placebo for 4 weeks as Cohort 5 and 6
Arm/Group | Multiple-dose (Cohort 5):0.3% SJP-0132 | Multiple-dose (Cohort 6):1% SJP-0132 | Multiple-dose (Cohort 5, 6):Placebo
Number analyzed (Participants) | 19 | 20 | 19
units on a scale | -34.2 (21.97) | -26.3 (22.00) | -29.8 (30.13)

7. Primary Outcome: Change From Baseline in Corneal Fluorescein Staining (CFS) Score at the Central Zone on Day 29
Description: Change from baseline of central zone CFS score at the central zone on Day 29. CFS score at the central zone ranged from 0 to 5, where '0' represents no fluorescein staining, and '5' represents severe staining on the cornea. The higher scores mean worse outcomes. Results from the study eye are reported.
Time Frame: Day 29
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Study eye
Arm/Group | Multiple-dose (Cohort 5) : 0.3% SJP-0132 | Multiple-dose (Cohort 6) : 1% SJP-0132 | Multiple-dose (Cohort 5, 6) : Placebo
Number analyzed (Participants) | 20 | 20 | 19
Number analyzed (Study eye) | 20 | 20 | 19
score on a scale | -1.1 (1.19) | -1.3 (1.08) | -1.2 (1.36)

8. Secondary Outcome: Change From Baseline in Eye Dryness Symptom by Visual Analog Scale (VAS) in Each Timepoints
Description: Visual analog scale (VAS): "0" mean none, and "100" mean the worst imaginable for the symptom question. Results from pre-dose are reported.
Time Frame: Day 29
Population: Full Analysis Set.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Multiple-dose (Cohort 5) : SJP-0132 Mid-High Dose: Multiple dose of Mid-High strength of SJP-0132 for 4 weeks as Cohort 5
- Multiple-dose (Cohort 6) : SJP-0132 High Dose: Multiple dose of High strength of SJP-0132 for 4 weeks as Cohort 6
Arm/Group | Multiple-dose (Cohort 5) : SJP-0132 Mid-High Dose | Multiple-dose (Cohort 6) : SJP-0132 High Dose | Multiple-dose (Cohort 5, 6) : Placebo
Number analyzed (Participants) | 20 | 20 | 20
score on a scale
  Day 2 | -14.3 (17.82) | -12.1 (17.92) | -8.0 (14.74)
  Day 8 | -29.7 (24.08) | -22.3 (21.33) | -24.2 (27.03)
  Day 15 | -30.1 (21.44) | -17.6 (21.03) | -22.8 (24.12)
  Day 22: number analyzed (Participants) | 19 | 20 | 19
  Day 22 | -30.3 (23.47) | -21.9 (22.21) | -28.9 (29.71)
  Day 29: number analyzed (Participants) | 20 | 20 | 19
  Day 29 | -34.6 (22.27) | -23.9 (22.46) | -26.8 (30.28)

9. Secondary Outcome: Change From Baseline in Corneal Fluorescein Staining (CFS) Score at Total Zone in Each Timepoints
Description: Change from baseline of CFS score at the total zone of pre-dose in each time point.
  Total zone means a summary of central, superior, inferior, nasal, and temporal zones.
  The range of the score in each zone is 0 to 5 points, and the total score is 25 points. The higher scores mean worse outcomes.
Time Frame: Day 8, 15, 22, 29
Population: Full Analysis Set.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Study eye
Arm/Group | Multiple-dose (Cohort 5) : 0.3% SJP-0132 | Multiple-dose (Cohort 6) : 1% SJP-0132 | Multiple-dose (Cohort 5, 6) : Placebo
Number analyzed (Participants) | 20 | 20 | 20
Number analyzed (Study eye) | 20 | 20 | 20
score on a scale
  Day 8 | -1.9 (4.84) | 0.6 (2.74) | -0.6 (2.96)
  Day 15 | -3.9 (3.92) | -0.2 (4.76) | -2.3 (5.70)
  Day 22: number analyzed (Participants) | 19 | 20 | 19
  Day 22: number analyzed (Study eye) | 19 | 20 | 19
  Day 22 | -4.4 (3.50) | 0.2 (5.16) | -1.4 (3.85)
  Day 29: number analyzed (Participants) | 20 | 20 | 19
  Day 29: number analyzed (Study eye) | 20 | 20 | 19
  Day 29 | -3.4 (3.82) | -1.8 (5.15) | -1.8 (4.94)

10. Secondary Outcome: Change From Baseline in Conjunctival Lissamine Green Staining (CLGS) Score at Total Zone in Each Timepoints
Description: The score in each zone is 0 to 5 points, and the maximum total score is 30 points. The higher scores mean worse outcomes. Results from the study eye are reported.
Time Frame: Day 8, 15, 22, 29
Population: Full Analysis Set.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Study eye
Arm/Group | Multiple-dose (Cohort 5) : 0.3% SJP-0132 | Multiple-dose (Cohort 6) : 1% SJP-0132 | Multiple-dose (Cohort 5, 6) : Placebo
Number analyzed (Participants) | 20 | 20 | 20
Number analyzed (Study eye) | 20 | 20 | 20
score on a scale
  Day 8 | 0.6 (5.25) | 1.7 (5.28) | 0.3 (3.80)
  Day 15 | 0.5 (5.66) | 2.1 (5.35) | 1.6 (3.93)
  Day 22: number analyzed (Participants) | 19 | 20 | 19
  Day 22: number analyzed (Study eye) | 19 | 20 | 19
  Day 22 | 0.5 (4.97) | 1.9 (4.15) | 1.8 (4.44)
  Day 29: number analyzed (Participants) | 20 | 20 | 19
  Day 29: number analyzed (Study eye) | 20 | 20 | 19
  Day 29 | 0.5 (5.95) | 1.4 (5.43) | 2.3 (4.26)

11. Secondary Outcome: Change From Baseline in Lid Wiper Epitheliopathy Score in Each Timepoints
Description: Lissamine green staining of the lid wiper was graded from 0 to 3. The higher scores mean worse outcomes. Results from the study eye are reported.
Time Frame: Day 8, 15, 22, 29
Population: Full Analysis Set.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Study eye
Groups:
- Multiple-dose (Cohort 6): 1% SJP-0132: Multiple dose of 1% SJP-0132 for 4 weeks as Cohort 6
Arm/Group | Multiple-dose (Cohort 5) : 0.3% SJP-0132 | Multiple-dose (Cohort 6): 1% SJP-0132 | Multiple-dose (Cohort 5, 6) : Placebo
Number analyzed (Participants) | 20 | 20 | 20
Number analyzed (Study eye) | 20 | 20 | 20
score on a scale
  Day 8 | -0.10 (0.620) | -0.33 (0.520) | -0.50 (0.973)
  Day 15 | 0.08 (0.799) | -0.40 (0.641) | -0.33 (0.963)
  Day 22: number analyzed (Participants) | 19 | 20 | 19
  Day 22: number analyzed (Study eye) | 19 | 20 | 19
  Day 22 | -0.13 (0.496) | -0.35 (0.630) | -0.18 (0.989)
  Day 29: number analyzed (Participants) | 20 | 20 | 19
  Day 29: number analyzed (Study eye) | 20 | 20 | 19
  Day 29 | -0.70 (1.081) | -0.43 (0.730) | -0.53 (0.993)

12. Secondary Outcome: Change From Baseline in Tear Film Break-up Time (TFBUT) in Each Timepoints
Description: Tear film break-up time is the time taken for the first dry spot to appear on the cornea after a complete blink.
Time Frame: Day 8, 15, 22, 29
Population: Full Analysis Set. One participant in placebo group was not completed the study.
Measure: Mean (Standard Deviation); unit: sec
Units Other Than Participants: Study eye
Arm/Group | Multiple-dose (Cohort 5) : 0.3% SJP-0132 | Multiple-dose (Cohort 6) : 1% SJP-0132 | Multiple-dose (Cohort 5, 6) : Placebo
Number analyzed (Participants) | 20 | 20 | 20
Number analyzed (Study eye) | 20 | 20 | 20
sec
  Day 8: number analyzed (Participants) | 20 | 20 | 19
  Day 8: number analyzed (Study eye) | 20 | 20 | 19
  Day 8 | 0.54 (2.580) | -0.04 (1.834) | 0.52 (2.024)
  Day 15 | 1.26 (2.848) | 0 (1.789) | -0.08 (2.755)
  Day 22: number analyzed (Participants) | 19 | 20 | 18
  Day 22: number analyzed (Study eye) | 19 | 20 | 18
  Day 22 | 0.98 (2.560) | -0.29 (1.178) | 0.89 (2.212)
  Day 29: number analyzed (Participants) | 20 | 20 | 19
  Day 29: number analyzed (Study eye) | 20 | 20 | 19
  Day 29 | 1.29 (3.435) | 0.32 (2.147) | 0.66 (1.720)

13. Secondary Outcome: Change From Baseline in Ocular Surface Disease Index (OSDI)
Description: The OSDI questionnaire consists of 12 questions regarding ocular symptoms, environmental triggers, and vision-related functioning. The participant was asked to rate each question using a 5-point scale (0 to 4), where 0 = none of the time; 1 = some of the time; 2 = half of the time; 3 = most of the time; and 4 = all of the time. The total OSDI was calculated from the raw scores of each of the 12 questions based on the formula: ([sum of scores for all questions answered] X 25)/([total number of questions answered]).
  The OSDI can range from 0 (normal) to 100 (abnormal).
Time Frame: Day 8, 15, 22, 29
Population: Full Analysis Set.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Multiple-dose (Cohort 5) : 0.3% SJP-0132 | Multiple-dose (Cohort 6) : 1% SJP-0132 | Multiple-dose (Cohort 5, 6) : Placebo
Number analyzed (Participants) | 20 | 20 | 20
score on a scale
  Day 8: number analyzed (Participants) | 19 | 20 | 20
  Day 8 | -24.19 (22.037) | -9.67 (19.494) | -28.17 (18.536)
  Day 15 | -22.94 (22.554) | -9.94 (20.342) | -23.91 (17.298)
  Day 22: number analyzed (Participants) | 19 | 20 | 19
  Day 22 | -24.02 (22.182) | -9.04 (20.266) | -22.21 (20.100)
  Day 29: number analyzed (Participants) | 20 | 20 | 19
  Day 29 | -24.38 (21.891) | -9.30 (22.785) | -23.54 (23.508)

14. Secondary Outcome: Change From Baseline in Dry Eye Questionnaire 5 (DEQ-5) Scores
Description: The participants rated the frequency on a scale of 0 (never) to 4 (constant) with which they have experienced 3 symptoms (watery eyes, discomfort and dryness). The participant was also asked to rate the intensity of discomfort and dryness on a scale of 0 (never have it) to 5 (very intense). Total DEQ-5 score was the sum of scores for frequency and intensity of dryness and discomfort plus frequency of watery eyes. Maximum score is 22.
  Higher scores mean a worse outcome.
Time Frame: Day 29
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Multiple-dose (Cohort 5) : 0.3% SJP-0132 | Multiple-dose (Cohort 6) : 1% SJP-0132 | Multiple-dose (Cohort 5, 6) : Placebo
Number analyzed (Participants) | 20 | 20 | 19
score on a scale | -6.0 (3.46) | -4.9 (4.00) | -3.6 (3.59)

15. Secondary Outcome: Change in Matrix Metalloproteinase-9 (MMP-9)
Description: Levels of the inflammatory marker Matrix Metalloproteinase-9 (MMP-9) were measured in each eye using InflammaDry. The test was recorded as either positive or negative. Results from the study eye are reported.
Time Frame: Day 29
Population: Full Analysis Set
Measure: Count of Units; unit: Study eye
Units Other Than Participants: Study eye
Arm/Group | Multiple-dose (Cohort 5) : 0.3% SJP-0132 | Multiple-dose (Cohort 6) : 1% SJP-0132 | Multiple-dose (Cohort 5, 6) : Placebo
Number analyzed (Participants) | 20 | 20 | 20
Number analyzed (Study eye) | 20 | 20 | 20
Study eye
  Baseline: Positive | 14 | 2 | 8
  Baseline: Negative | 6 | 18 | 12
  Baseline: Missing | 0 | 0 | 0
  Day 29: Positive | 2 | 4 | 7
  Day 29: Negative | 18 | 16 | 12
  Day 29: Missing | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: Day 2 for cohort 1-4, Day 29 for cohort 5-6
Description: Adverse events are reported as Treatment-Emergent Adverse Events (TEAEs), which are defined as any event not present before exposure to the study drug or any event already presented that worsened in either intensity or frequency after exposure to the study drug.
Groups:
- Single-dose (Cohort 1) : SJP-0132 Low Dose: Single dose of Low strength of SJP-0132 as Cohort 1
- Single-dose (Cohort 2) : SJP-0132 Mid-Low Dose: Single dose of Mid-Low strength of SJP-0132 as Cohort 2
- Single-dose (Cohort 3) : SJP-0132 Mid-High Dose: Single dose of Mid-High strength of SJP-0132 as Cohort 3
- Single-dose (Cohort 4) : SJP-0132 High Dose: Single dose of High strength of SJP-0132 as Cohort 4
Arm/Group | Single-dose (Cohort 1) : SJP-0132 Low Dose | Single-dose (Cohort 2) : SJP-0132 Mid-Low Dose | Single-dose (Cohort 3) : SJP-0132 Mid-High Dose | Single-dose (Cohort 4) : SJP-0132 High Dose | Single-dose (Cohort 1-4) : Placebo | Multiple-dose (Cohort 5) : SJP-0132 Mid-High Dose | Multiple-dose (Cohort 6) : SJP-0132 High Dose | Multiple-dose (Cohort 5, 6) : Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/5 | 0/4 | 0/8 | 0/20 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/5 | 0/4 | 0/8 | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 2/5 | 0/4 | 0/8 | 1/20 | 5/20 | 7/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single-dose (Cohort 1) : SJP-0132 Low Dose (N=6) | Single-dose (Cohort 2) : SJP-0132 Mid-Low Dose (N=6) | Single-dose (Cohort 3) : SJP-0132 Mid-High Dose (N=5) | Single-dose (Cohort 4) : SJP-0132 High Dose (N=4) | Single-dose (Cohort 1-4) : Placebo (N=8) | Multiple-dose (Cohort 5) : SJP-0132 Mid-High Dose (N=20) | Multiple-dose (Cohort 6) : SJP-0132 High Dose (N=20) | Multiple-dose (Cohort 5, 6) : Placebo (N=20)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Conjunctival hemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sensitive skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
All of the efficacy and safety measurements applied in this study are widely used and generally recognized as reliable, accurate, and relevant.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-12): https://cdn.clinicaltrials.gov/large-docs/22/NCT04139122/Prot_SAP_001.pdf